CLINICAL TRIAL: NCT02939417
Title: One Year Clinical Evaluation of E.Max Laminate Veneers With and Without Using Grape Seed Extract as a Natural Collagen Cross-linking Agent Before Bonding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marwa Salem (Other)
Responsible Party: Sponsor-Investigator, Marwa Salem, Marwa Salem, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBC-CU-201610168
Record Dates: First submitted 2016-10-17; First posted 2016-10-20 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Retention & Fracture of Emax Laminate Veneers
Keywords: Laminate veneers; Grape seed extract; Emax; collagen cross-linking agent
MeSH Terms: interventions — Grape Seed Extract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- using grape seed extract (Experimental): Grape seed extract as collagen cross-linking agent
  Interventions: Other: Grape seed extract
- without uing grape seed extract (Active Comparator)
  Interventions: Other: Grape seed extract

INTERVENTIONS:
Other: Grape seed extract — Grape seed extract - collagen cross-linking agent

SUMMARY:
The aim of this study is to evaluate the clinical performance of E-max veneers cemented with and without using grape seed extract before bonding.

DETAILED DESCRIPTION:
Justification for undertaking the trial:

Ceramic veneers have become a popular dental procedure since its introduction because they provide excellent esthetics.1 Achieving the good esthetic results especially with ceramic veneers is probably the most challenging task encountered by dental practitioners and ceramist today. Ceramic veneers are indicated for teeth with moderate discoloration, restoration of traumatized, fractured, worn dentition and abnormal tooth anatomy.2 Many factors affect the long term success of ceramic laminate veneers. The most repeated failure patterns associated with ceramic laminate veneer were fractures, microleakage, colour change and detachment of restoration.3 The main reasons for failure were large marginal defect and fractures.4 The clinical performance of ceramic veneer has shown that the estimated survival rate for the teeth prepared with butt joint design are higher than for the teeth prepared with palatal chamfer design.5 The bonding technique, which is a time-consuming and technique sensitive procedure, is a key to the long-term success of these types of restorations. The strength and the durability of the bond between the porcelain, the luting cement and the enamel/dentin interface play an important role in the outcome of ceramic veneers, particularly when dentin is involved. 6

Expected benefits for the patient

1. Achieving a more predictable esthetic restoration while being conservative. 2. Increasing the long term prognosis of the restoration. Expected benefits for the clinician

1. Enriching the professional skills of the dentist with a new material to improve the clinical performance of the restoration.
2. Improving the confidence in the patient-dentist relationship.

Explanation for Choice of Comparators Resin cements are generally used for the bonding of all ceramic restorations since they provide adequate aesthetics, low solubility in oral environment, high bond strength to tooth structures, superior mechanical properties and support for ceramic.7 Since their retention relies solely on adhesion, durable adhesion of resin luting cements to both the enamel/dentin and the cementation surface of the ceramic is crucial. Luting cements used in conjunction with phosphoric acid etching followed by adhesive application on enamel show reliable adhesion.8 By studying the effect of incorporation of natural cross-linkers into the primer of a self-etching adhesive on resin-dentine bond strength, it had a positive influence on the immediate μTBS (micro tensile bond strength) and mechanical properties of the bonded interface.9

Statement of problem:

Ceramic veneers have become a popular dental procedure since its introduction because they provide excellent esthetics while being conservative. However, high failure rates of PLVs have been attributed to the exposure of dentin surface during preparation which greatly decrease the bonding strength at the dentin-cement interface. Natural and synthetic cross-linking agents have been introduced to restore dentin function, enhance bonding strength as well as positively affect the remineralization process in artificial roots. They have the ability to enhance the mechanical properties and stability of dentin matrix by the use of PA-rich collagen cross-linkers most likely due to the formation of a PA-collagen complex.10

Research hypothesis The null hypothesis of the study that there won't be a difference in the clinical performance & adhesion of laminate veneers after application of grape seed extract before bonding.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 20-40 years old, able to read and sign the informed consent document.
2. Patients having teeth with exposed dentin surface limited to cervical third.
3. Patients, healthy physically and psychologically, able to tolerate conventional restorative procedures.
4. Patients don't have active periodontal or pulpal diseases and have teeth with good restorations.
5. Patients with normal occlusion.
6. Patients with teeth problems indicated for laminate veneer (e.g. discoloration, mild malposition, fracture not involving more than 50% enamel loss, ….)
7. Patients willing to return for follow-up examination and evaluation.

Exclusion Criteria:

1. Patients in the growth stage with partially erupted teeth.
2. Patients with fractured teeth with more than 50% enamel loss.
3. Patients with poor oral hygiene and lack of motivation.
4. Pregnant women.
5. Patients with abnormal occlusion (eg. edge to edge, deep bite, …)
6. Patients with parafunctional habits (eg. Bruxism, biting on hard objects, …)
7. Patients with endodontically treated teeth.
8. Lack of opposite occluding dentition in the area intended for restoration.
9. Psychiatric problems or unrealistic expectations.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Retention of laminate veneers | 1 year
  using USPHS criteria for clinical evaluation
Fracture of laminate veneers | 1 year
  using USPHS criteria for clinical evaluation
Marginal adaptation of laminate veneers | 1 year
  using USPHS criteria for clinical evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Heba Hamza, Professor, Study Director — Faculty of Oral and Dental Medicine- Cairo University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Prasanth, V., Harshakumar, K., Lylajam, S., K, C. N. & Sreelal, T. Relation between fracture load and tooth preparation of ceramic veneers - an in vitro study. Heal. Sci. 2, 1-11 (2013).
- [Background] Jankar AS, Kale Y, Kangane S, Ambekar A, Sinha M, Chaware S. Comparative evaluation of fracture resistance of Ceramic Veneer with three different incisal design preparations - An In-vitro Study. J Int Oral Health. 2014 Feb;6(1):48-54. Epub 2014 Feb 26. PMID 24653603
- [Background] Alghazzawi TF, Lemons J, Liu PR, Essig ME, Janowski GM. The failure load of CAD/CAM generated zirconia and glass-ceramic laminate veneers with different preparation designs. J Prosthet Dent. 2012 Dec;108(6):386-93. doi: 10.1016/S0022-3913(12)60198-X. PMID 23217471
- [Background] Sadighpour L, Geramipanah F, Allahyari S, Fallahi Sichani B, Kharazi Fard MJ. In vitro evaluation of the fracture resistance and microleakage of porcelain laminate veneers bonded to teeth with composite fillings after cyclic loading. J Adv Prosthodont. 2014 Aug;6(4):278-84. doi: 10.4047/jap.2014.6.4.278. Epub 2014 Aug 14. PMID 25177471
- [Background] da Costa DC, Coutinho M, de Sousa AS, Ennes JP. A meta-analysis of the most indicated preparation design for porcelain laminate veneers. J Adhes Dent. 2013 Jun;15(3):215-20. doi: 10.3290/j.jad.a29587. PMID 23593640
- [Background] Ibarra G, Johnson GH, Geurtsen W, Vargas MA. Microleakage of porcelain veneer restorations bonded to enamel and dentin with a new self-adhesive resin-based dental cement. Dent Mater. 2007 Feb;23(2):218-25. doi: 10.1016/j.dental.2006.01.013. Epub 2006 Feb 24. PMID 16499961
- [Background] Souza, P. & Lopes, L. G. Influence of the Resin Cement Color on the Shade of Porcelain Veneers After Accelerated Artificial Aging Influência da Cor do Cimento Resinoso na Tonalidade de Facetas de Porcelana Após Envelhecimento Artificial Acelerado. 21, (faculty of oral and dental medicine of cairo university, 2013).
- [Background] Gresnigt MM, Kalk W, Ozcan M. Clinical longevity of ceramic laminate veneers bonded to teeth with and without existing composite restorations up to 40 months. Clin Oral Investig. 2013 Apr;17(3):823-32. doi: 10.1007/s00784-012-0790-5. Epub 2012 Jul 21. PMID 22821429
- [Background] Islam S, Hiraishi N, Nassar M, Yiu C, Otsuki M, Tagami J. Effect of natural cross-linkers incorporation in a self-etching primer on dentine bond strength. J Dent. 2012 Dec;40(12):1052-9. doi: 10.1016/j.jdent.2012.08.015. Epub 2012 Sep 11. PMID 22982944
- [Background] Castellan CS, Pereira PN, Grande RH, Bedran-Russo AK. Mechanical characterization of proanthocyanidin-dentin matrix interaction. Dent Mater. 2010 Oct;26(10):968-73. doi: 10.1016/j.dental.2010.06.001. Epub 2010 Jul 21. PMID 20650510